CLINICAL TRIAL: NCT05113498
Title: The Influence of the Microbiome on the Pharmacokinetics of Flavan-3-ols After Acute Consumption in Healthy Young Male Participants
Brief Title: The Influence of the Microbiome on the Pharmacokinetics of Flavan-3-ols
Acronym: PhTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC-09585
Record Dates: First submitted 2021-10-15; First posted 2021-11-09 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Diet Modification
Keywords: Valerolactones; (-)-Epicatechin; Microbiota; Pharmacokinetics; Interindividual differences; Q-TOF-LC-MS
MeSH Terms: interventions — Catechin

STUDY DESIGN:
Intervention Model Description: Single-dose study where all participants consume one epicatechin supplement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (-)-Epicatechin (Experimental): (-)-Epicatechin supplementation
  Interventions: Dietary Supplement: (-)-Epicatechin

INTERVENTIONS:
Dietary Supplement: (-)-Epicatechin — Administration of a capsule with 150 mg of pure (-)-epicatechin after 48h low-flavanol diet.

SUMMARY:
Cocoa beans are of major interest due to their various beneficial health effects, indicated to be caused by its cocoa flavan-3-ols. (-)-Epicatechin is the most abundant flavan-3-ol in these cocoa beans. Its metabolization in the colon results in bioactive valerolactone and valeric acid metabolites and derivatives after phase II metabolism. Interindividual differences in health effects following (-)-epicatechin consumption are observed, which are suggested to be caused by large interindividual differences in bioavailable metabolite concentrations. As the colonic microbiota is responsible for the metabolization of ~70% of total (-)-epicatechin intake, and ~42% of total (-)-epicatechin intake leads to valerolactone and valeric acid metabolites, it is hypothesized that the large interindividual variation in microbial gut composition is responsible for the heterogeneity in metabolite concentration and in its subsequent health effects. Furthermore, individuals can be stratified into two pharmacotypes, slow and fast microbial metabolizers, which can produce metabolites at different rates.

The aim of this single-arm study is to investigate if the microbial composition in the gut determines the rate and extent of metabolization, following an acute consumption of about 160mg of pure (-)-epicatechin. The pharmacokinetics of the (-)-epicatechin metabolites will be followed in plasma over 48h with a focus on the first fifteen hours and potentially in urine over 24h. Valerolactone and valeric acid metabolite profiles in plasma and urine will be obtained by Q-TOF-LC-MS. The microbial fingerprint of each individual will be obtained via DNA extraction, flow cytometry and 16s rRNA sequencing of fecal samples.

DETAILED DESCRIPTION:
The aim of this study is to investigate if the microbial composition in the gut can determine the rate and extent of valerolactone and valeric acid production following an acute consumption of 160mg of pure (-)-epicatechin. The gut microbial composition of each participant will be linked with its metabolite plasma profile to investigate if the large interindividual variation in metabolite formation can be explained by the variation in microbial composition in the colon. This knowledge might contribute to a better understanding of the correlation between epicatechin intake and its observed beneficial, but at the same time very variable health effects.

This single-arm trial lasts a total of five days, with one day (day 3) on site at the laboratory (UZ Ghent, Department of Rehabilitation Sciences). Two days prior to the test day, subjects will be instructed to follow a low-flavan-3-ol diet for the next five days, until 48h after the supplement intake, to establish a low dietary background of flavan-3-ols. A list of restrictions on foods and beverages rich in flavan-3-ols, such as chocolate, tea, red wine and some fruit and vegetables, will be provided. Moreover, a standardized flavan-3-ol-free meal and snack will be provided to consume the evening prior to the test day, together with at least 0.5L of water. One day prior to the test day, each participant will collect a stool sample for the determination of their microbial fingerprint. Stool collection material will be provided to the subjects on beforehand. In addition, no strenuous exercise can be performed on this day.

On the test day, participants arrive at the laboratory around 8am after an overnight fast of minimum 8h and maximum 14h. This day lasts approximately 15h, until 11pm. First, a questionnaire will be completed to evaluate compliance with the instructed diet and to check the general well-being of the participants. Second, a medical doctor will insert a catheter in the median cubital vein in the forearm, after which a first blood sample will be drawn. Third, participants will be asked to empty the bladder, have breakfast and take the epicatechin supplement within ten minutes after breakfast. Standardized flavan-3-ol-free breakfast, lunch, dinner and three snacks will be offered at scheduled time points throughout the day. Water is ad libitum with a minimum of 1.5L. Lastly, a food frequency questionnaire will be completed.

Each hour after supplement intake, venous blood will be drawn in vacutainers until fifteen samples of 4mL are collected (0h-14h). On time points 0, 2, 6, 8 and 12h, additional blood samples will be drawn in serum vacutainers. Urine will be pooled in three timeframes (0-6h, 6-12h and 12-24h). When all blood samples are collected, the catheter will be removed and a questionnaire will be completed to evaluate the test day and well-being of the participants. On each of the two following mornings (24h and 48h), one additional blood sample will be taken after an overnight fast. The pooled urine (12-24h) will be collected 24h after supplement intake. Some participants will also conduct this trial without the (-)-epicatechin supplement to verify the effectiveness of the flavan-3-ol-free diet .

Valerolactone and valeric acid metabolite profiles will be obtained by Quadrupole Time of Flight Liquid chromatography-mass spectrometry (Q-TOF-LC-MS). The microbial fingerprint of each individual will be obtained via DNA extraction, flow cytometry and 16s rRNA sequencing of fecal samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Stable diet
* Stable exercise regimen

Exclusion Criteria:

* The use of antibiotics, pre- and probiotics in the last six months
* The use of chronic medication
* The use of any medication in the last 2 weeks
* Diarrhea in last 2 weeks
* Recent blood donations
* Vegan or vegetarian diets
* Smoking
* Chronic pathology or gastrointestinal disorders

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Assessing the formation of phase II valerolactone and valeric acid metabolites over time in blood. | 48 hours
  Assessing the concentration of colonic valerolactone and valeric acid metabolites over time in blood by Q-TOF-LC-MS, after the consumption of 160g pure (-)-epicatechin, to identify poor and extensive metabolizers.
Identification of the bacteria on genus level in fecal samples of participants. | Baseline
  All bacteria in the fecal samples of participants will be identified by 16S rRNA gene-based analysis on genus level.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Rietzschel, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No
After publication (or during the review process) of the scientific paper individual data will be made available upon request to the corresponding author. Data that allows for identification of the participants will never be provided.

REFERENCES:
- [Background] Mena P, Bresciani L, Brindani N, Ludwig IA, Pereira-Caro G, Angelino D, Llorach R, Calani L, Brighenti F, Clifford MN, Gill CIR, Crozier A, Curti C, Del Rio D. Phenyl-gamma-valerolactones and phenylvaleric acids, the main colonic metabolites of flavan-3-ols: synthesis, analysis, bioavailability, and bioactivity. Nat Prod Rep. 2019 May 22;36(5):714-752. doi: 10.1039/c8np00062j. PMID 30468210